CLINICAL TRIAL: NCT04256213
Title: A Multicenter, Pilot Study Evaluating Immune Impact and Safety of Nivolumab in Combination with Ipilimumab (immune Combination) Before Initial RT-CT Treatment for Cervix Cancer.: the French GINECO - COLIBRI Study
Brief Title: COL Immunotherapy Before Radiochimio + Ipilimumab
Acronym: COLIBRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GINECO-CE108b; 2019-002271-34 (EudraCT Number)
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Cervix Cancer
Keywords: Cervix cancer; Immune combination
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab + Ipilimumab (Experimental)
  Interventions: Drug: Nivolumab and Ipilimumab

INTERVENTIONS:
Drug: Nivolumab and Ipilimumab — Nivolumab, IV D1C1 and D15C1 (before RT-CT) at 3 mg/kg Every 28 days at 480 mg during 6 months after RT-CT
  Ipilimumab, 1 mg/kg, IV D1C1 (before RT-CT)

SUMMARY:
This is a multicenter, single arm pilot study evaluating the biological impact of "Nivolumab + Ipilimumab" in patients with cervical squamous cell carcinoma requiring RT-CT as initial therapy

DETAILED DESCRIPTION:
The aim of COLIBRI is to evaluate the evolution of the CD8+/FOXP3+ ratio of lymphocytes in pre- versus post-treatment biopsies in patients treated with a combination of Nivolumab and Ipilimumab in a pilot study, just before starting standard RT-CT.

The study will also assess tolerability, Objective Response Rate, clinical activity and biological (dynamic) changes of the immune micro environment

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed diagnosis of cervical squamous cell carcinoma stage IB3 to IVA, (FIGO 2018)

* Patients requiring RT-CT therapy as standard of care
* Age ≥18
* Patient accepting to undergo a new cervix biopsy
* Adequate marrow function:

  * White blood cell (WBC) >2000/mm3 (stable off any growth factor within 4 weeks of first study drug administration)
  * Neutrophils >1500/ mm3 (stable off any growth factor within 4 weeks of first study drug administration)
  * Platelets > 100× 103/mm3 (transfusion to achieve this level is not permitted within 2 weeks of first study drug administration)
  * Hemoglobin > 8 g/dL (transfusion to achieve this level is not permitted within 2 weeks of first study drug administration)
* Adequate other organ functions:

  * ALT and AST < 3× institutional ULN
  * Total bilirubin < 1.5× institutional ULN (except subjects with Gilbert's Syndrome who must have normal direct bilirubin)
  * Normal thyroid function, subclinical hypothyroidism (thyroid-stimulating hormone [TSH] < 10 mIU/mL) or have controlled hypothyroidism on appropriate thyroid supplementation
  * Serum creatinine < 2× ULN or creatinine clearance (CrCl) > 40 mL/min (measured using the Cockcroft-Gault formula or the MDRD formula for patients older than 65 years-old
* General Health as evidenced by PS ≤2
* Covered by a medical insurance
* Signed and dated informed consent form prior to any study-specific procedure.
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Women of childbearing potential must have a negative serum or urine pregnancy test For females of reproductive potential: use of highly effective contraception and for at least 5 months after administration of the last dose of nivolumab. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmeno-pausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries, fallopian tubes, and/or uterus).
* All subjects must consent to allow the acquisition of blood samples, FFPE tumor tissue, either a block or 15 to 20 unstained slides, and fresh tumor for performance of correlative studies.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Patient concurrently using other approved or investigational antineoplastic agents.
* Patient candidate for neo adjuvant CT before RT-CT
* Any contraindication to nivolumab or ipilimumab treatments as per Nivolumab and Ipilimumab Investigator's Brochure
* Prior therapy with an immune checkpoint inhibitor
* Prior history of other malignancies other than study disease (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the patient has been free of the disease for at least 3 years.
* Immune-deficient status (patients with HIV, immunosuppressive treatment, haematological malignancies, and previous organ transplantation)
* History of any chronic hepatitis as evidenced by:

  * Positive test for hepatitis B surface antigen
  * Positive test for qualitative hepatitis C viral load (by polymerase chain reaction [PCR])

Note: Subjects with positive hepatitis C antibody and negative quantitative hepatitis C by PCR are eligible. History of resolved hepatitis A virus infection is not an exclusion criterion

* Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

  * Myocardial infarction or stroke/transient ischemic attack within the past 6 months
  * Uncontrolled angina within the past 3 months
  * History of other clinically significant heart disease (eg, cardiomyopathy, congestive heart failure with New York Heart Association functional classification III-IV, pericarditis, significant pericardial effusion, or myocarditis)
  * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
  * QT interval corrected for heart rate using Fridericia's formula (QTcF) prolongation > 480 msec
  * Cardiovascular disease-related requirement for daily supplemental oxygen therapy
* Subjects with known or suspected CNS metastases, untreated CNS metastases, are excluded.

Note: However, subjects with controlled brain metastases will be allowed to enroll. Controlled brain metastases are defined as no radiographic progression for at least 4 weeks following radiation and/or surgical treatment (or 4 weeks of observation if no intervention is clinically indicated), and off of steroids for at least 2 weeks, and no new or progressive neurological signs and symptoms.

• Patients requiring concomitant treatment with therapeutic doses of anticoagulants will not be eligible for this clinical trial.

Note: Patients treated with low dose of anticoagulants for thrombo-embolic events prophylaxis are allowed.

• Any major surgery within 4 weeks of study drug administration. Subjects must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before the first dose of study drug.

Note: Pelvic and aortic dissection is not considered as traumatic surgery, and therefore can be performed if clinically indicated.

* Subjects with active, known or suspected autoimmune disease. Note: Subjects with skin disorders (such as vitiligo, psoriasis or alopecia), type I diabetes mellitus, hypothyroidism only requiring hormone replacement or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration.

Note: Inhaled or topical steroids, and adrenal replacement doses are permitted in the absence of active autoimmune disease.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2024-08-04 (Actual)

PRIMARY OUTCOMES:
CD8+/FOXP3+ relative change of lymphocytes from pre to post treatment biopsies | Baseline, before RT-CT

SECONDARY OUTCOMES:
Adverse events | Up to 100-days after end of treatment or until initiation of alternative cancer therapy
  Assessed by CTCAE 4.03
Objective Response Rate | 1week before RT-CT, 4 weeks after RT-CT
Progression Free Survival | 1 year
Overall Survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle RAY-COQUARD, MD, PhD, Principal Investigator — Centre Leon Berard
Locations (8):
- France (8):
  - Centre François Baclesse, Caen
  - Centre Léon Bérard, Lyon
  - Groupe Hospitalier Diaconesses - Croix Saint-Simon, Paris
  - Institut Curie, Paris
  - Centre Armoricain de Radiothérapie, Imagerie médicale et Oncologie, CARIO-HPCA, Plérin
  - Institut Jean Godinot, Reims
  - Institut Claudius Regaud IUCT-O, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy